CLINICAL TRIAL: NCT04385316
Title: Clinical Study of Gastric Cancer, Colorectal Cancer and Bladder Cancer Based on Liquid Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-SR-369
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Gastric Cancer; Colorectal Cancer; Bladder Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gastric Cancer
  Interventions: Diagnostic Test: DNA extraction of samples and high-throughput sequencing of small panels
- Colorectal Cancer
  Interventions: Diagnostic Test: DNA extraction of samples and high-throughput sequencing of small panels
- Bladder Cancer
  Interventions: Diagnostic Test: DNA extraction of samples and high-throughput sequencing of small panels

INTERVENTIONS:
Diagnostic Test: DNA extraction of samples and high-throughput sequencing of small panels — DNA extraction of gastric tumor tissues and high-throughput sequencing of small panels were performed, and the relationship between the mutation spectrum of each sample and the corresponding patient clinical data (staging) was analyzed.
  DNA extraction of tumer tissue samples and blood sample and high-throughput sequencing of small panels,DNA extraction and small panel sequencing were performed for the two types of samples of the patients respectively, and the DNA sequencing results of the two types of samples were compared, and the clinical data of the corresponding patients were referenced to evaluate the consistency of the results of peripheral blood ctDNA and tissue gDNA for the gene detection of gastric tumor.
  Groups: Gastric Cancer
Diagnostic Test: DNA extraction of samples and high-throughput sequencing of small panels — DNA extraction of colorectal tumor tissues and high-throughput sequencing of small panels were performed, and the relationship between the mutation spectrum of each sample and the corresponding patient clinical data (staging) was analyzed.
  DNA extraction of tumer tissue samples and blood sample and high-throughput sequencing of small panels,DNA extraction and small panel sequencing were performed for the two types of samples of the patients respectively, and the DNA sequencing results of the two types of samples were compared, and the clinical data of the corresponding patients were referenced to evaluate the consistency of the results of peripheral blood ctDNA and tissue gDNA for the gene detection of colorectal tumor.
  Groups: Colorectal Cancer
Diagnostic Test: DNA extraction of samples and high-throughput sequencing of small panels — DNA extraction of bladder tumor tissues and high-throughput sequencing of small panels were performed, and the relationship between the mutation spectrum of each sample and the corresponding patient clinical data (staging) was analyzed.
  DNA extraction of tumer tissue samples ,urine sample，blood sample and high-throughput sequencing of small panels,DNA extraction and small panel sequencing were performed for the three types of samples of the patients respectively, and the DNA sequencing results of the three types of samples were compared, and the clinical data of the corresponding patients were referenced to evaluate the consistency of the results of peripheral blood ctDNA ,urine ctDNAand tissue gDNA for the gene detection of bladder tumor.
  Groups: Bladder Cancer

SUMMARY:
Gastric cancer and colorectal cancer are common gastrointestinal malignancies in the world.Early cancer generally has no obvious symptoms. Endoscopy is the "gold standard"for the diagnosis of gastric cancer and colorectal cancer.gastric cancer and colorectal cancer treatment mainly includes surgery and medication.Compared with traditional diagnosis and treatment methods, the application of gene detection technology, especially high-throughput sequencing technology (NGS) in tumor diagnosis and treatment, performs multi-dimensional and multi-target detection of cancer-related genes, which can quickly and accurately determine the target gene mutations Morphology and expression differences, so as to provide personalized guidance to patients in terms of medication, treatment or prognosis evaluation, which can save a lot of time and treatment costs, and improve the overall treatment effect and patient quality of life.

Cystoscopy and biopsy sampling pathological testing are the gold standard for bladder cancer diagnosis, and have been widely used in clinical diagnosis and prognosis judgment. However, cystoscopy is cumbersome, expensive, and often causes pain to the patients under test. At present, the main clinical non-invasive detection technique for bladder cancer is still the cytological examination of urinary tract bladder cells in urine, and its sensitivity and specificity are not good, especially for the diagnosis of early lower grade bladder cancer.For bladder cancer, tumor tissue (puncture biopsy or surgical resection) DNA, urine ctDNA, urinary tract exfoliated cell DNA and peripheral blood ctDNA can be used for genetic testing, but the consistency of the genetic testing results of these four types of samples has not been verified, especially There is no systematic evaluation of the guidance effect of non-invasive gene detection of free tumor DNA and urinary tract shed cell DNA in the diagnosis and treatment of bladder cancer.The corresponding relationship between the significant mutation genes contained in the DNA derived from bladder urinary tract cancer and the various types and stages of bladder cancer is not clear.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for gastric tumor, colorectal tumor or bladder tumor resection Signed informed consent

Exclusion Criteria:

* the vital signs are not stable unconscious unwilling to cooperate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastric cancer, colorectal cancer or bladder cancer patients in Jiangsu Provincial People's Hospital
Sampling Method: Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
DNA extraction of tumer tissue samples and high-throughput sequencing | 2019.9-2019.6
  Preliminary exploration of tumor related mutation spectrum in different patients by gene sequencing

SECONDARY OUTCOMES:
DNA extraction of tumer tissue samples, blood tissue and urine samples and high-throughput sequencing | 2020.7-2020.12
  To evaluate the consistency of peripheral blood ctDNA and tissue gDNA in gene detection of gastric cancer and colorectal cancer.
  To evaluate the consistency of peripheral blood ctDNA , urine ctDNA and tissue gDNA in gene detection of bladder cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical Universit, Nanjing, Jiangsu, China